CLINICAL TRIAL: NCT05323604
Title: Impact of Sarcopenia on Post-operative Course for Cancer Patients Operated of Colorectal Surgery Using a Simple Measurement Method of the Psoas Muscle Surface Area
Brief Title: Impact of Sarcopenia Using an Easy Psoas Area Measurement
Acronym: ISEPAM
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD3021
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-04

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; colorectal neoplasm; colorectal surgery; psoas muscles
MeSH Terms: conditions — Sarcopenia; Colorectal Neoplasms | interventions — Colectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Colectomy with anastomosis of any type: Patient with colonic resection followed by ileocolic, or colo colic, or colorectal, or coloanal anastomosis for cancer by laparoscopy or laparotomy
  Interventions: Other: Colectomy with anastomosis of any type

INTERVENTIONS:
Other: Colectomy with anastomosis of any type — Patient with colonic resection followed by ileocolic, or colo colic, or colorectal, or coloanal anastomosis for cancer by laparoscopy or laparotomy

SUMMARY:
The purpose of this study is to compare the post-operative course in patients suffering from sarcopenia who had colorectal surgery for cancer. Our primary outcome is the comparaison of the length of hospital stay in sarcopenic and non sarcopenic patients.

DETAILED DESCRIPTION:
Sarcopenia is the loss of muscle mass that occurs usually with aging, but it may have multiple contributing factors, especially related to chronic diseases such as colorectal cancer.

When present, sarcopenia is predictive of poor post-operative course. The identification of sarcopenia needs either the identification of low muscle strength, low muscle quantity/quality, or finally a low physical performance.

Multiple clinical, biological or radiological tools were proposed. Our purpose is to compare the post-operative outcome of sarcopenic and non sarcopenic patients using a simple, available, reproducible and rapid radiological method, which will help the healthcare professionals to rapidly identify high risk patients for possible complicated and long post-operative course allowing them to take appropriate perioperative measures to reduce the risks.

ELIGIBILITY:
Inclusion Criteria:

* Patient operated on for colectomy or proctectomy with restoration of continuity for colorectal cancer between 1 January 2020 and 31 December 2021
* Patient who had a CT scan in the 2 months prior surgery
* Patient aged 18 years or older

Exclusion Criteria:

* Patients with inflammatory bowel disease (Crohn disease, haemorrhagic rectocolitis)
* Patients with neuromuscular pathology affecting their mobility
* Patients who were diagnosed positif to SARS COV 2 before or during hospitalisation
* Patients who refuse the collection of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from sarcopenia who had colorectal surgery for cancer.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the average postoperative length of stay in sacopenic and non-sarcopenic patients | Until discharge from hospital, an average of 30 days
  Comparison of the number of post-operative hospital days between the two groups

SECONDARY OUTCOMES:
Comparison between complication rate in sarcopenic and non sarcopenic patients | At the end of the 30 post-operative days
  Measurement of the complication rate according to the Clavien Dindo score (relevant score if greater than or equal to 2, considered severe complication if greater than or equal to 3) between the two groups
Assessment of re-hospitalization rate between sarcopenic and non sarcopenic patients | At the end of the 30 post-operative days
  Evaluation of the number of hospitalizations of more than 24 hours at 30 days after the operation between the two groups
Comparison of the transfer rate to rehabilitation or nursing home center between sarcopenic and non sarcopenic patients | At the end of the 30 post-operative days
  Evaluation of the number of transfer to rehabilitation or nursing home center at 30 days after the operation between the two groups
Comparison of the length of stay in the rehabilitation center for sarcopenic and non sarcopenic transferred patients | At the end of the 30 post-operative days
  Comparison of the number of hospital days for transferred patients between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Hicham El Masri, Principal Investigator — Hospital René Dubos
Locations (1):
- Centre Hospitalier René Dubos, Pontoise, France

IPD SHARING:
Plan to Share IPD: No